CLINICAL TRIAL: NCT00845637
Title: Effect of the Oral Administration of Eggplant Extract Capsules on Lipid Profile During Fasting and Postprandial Period: a Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Effect of Eggplant Extract on Lipid Profile During Fasting and Postprandial Period
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Paulo Dornelles Picon, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04004
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Dyslipidemia
Keywords: eggplant; dyslipidemia; postprandial lipemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eggplant extract (Active Comparator)
  Interventions: Drug: Eggplant extract
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eggplant extract — Dry eggplant extract in two 450mg capsules, twice a day (before the main meals) for fourteen days.
  Arms: Eggplant extract
Drug: Placebo — Placebo in two 450mg capsules, twice a day (before the main meals) for fourteen days.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the effect of eggplant extract capsules on the lipid profile of healthy individuals after an oral lipid overload test in a randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Dry eggplant extract(Solanum melongena) has been used by the population as an alternative treatment for dyslipidemia. It is a vegetable rich in flavonoids, which are polyphenol anti-oxidants found in foods. Studies suggest an inverse relationship between the ingestion of foods rich in flavonoids and mortality from coronary artery disease. The aim of this study was to assess the effect of administering eggplant extract capsules on the lipid profile of healthy individuals after an oral lipid overload test.

Participants underwent a baseline clinical evaluation conducted by a doctor, who assessed whether the volunteer was apt to participate in the study. Diabetics, smokers and users of hypolipidemic medication were excluded. After signing an informed consent form, 59 healthy volunteers of both genders were randomized to take either capsules containing 450 mg of dry eggplant extract or placebo. Both interventions were administered in quantities of two capsules, twice a day, for 14 days, and both patient and doctor were unaware of the drug in use.

The main outcome measure was lipid profile, which was checked during fasting on days 0 and 14, and also during postprandial period on the 14th day, when participants underwent a lipid overload test immediately after ingesting 900 mg of eggplant extract or placebo, as per prior randomization. The nutritional analysis of the meal contained 361 kcal and 22.5g of total fat, 14.5 g of which was saturated and 251mg of cholesterol. Laboratory exams were taken (total cholesterol, triglycerides, HDL-C). LDL-C was calculated according to the Friedewald formula: LDL-C = CT - HDL-C - TG/5. The nutritional value of food records was conducted with the help of Diet Win for Windows nutritional evaluation software.

Anthropometric evaluation was also performed, including body weight, height and abdominal circumference, at baseline and on day 14, by the same investigator, blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Baseline clinical evaluation conducted by a doctor
* Informed consent form

Exclusion Criteria:

* Diabetes Mellitus
* Smoking
* Use of hypolipidemic medication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Lipid profile | Before treatment and twice on the fouteenth day, before and 2 hours after lipid overload test

SECONDARY OUTCOMES:
Anthropometric measures | Before treatment and on day fourteen

CONTACTS AND LOCATIONS:
Overall Officials: Paulo D Picon, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil